CLINICAL TRIAL: NCT02979392
Title: A Prospective, Open-label, Dose Escalation (Part A), Cohort Expansion (Part B) Phase I Study to Investigate the Safety and to Determine Maximum Tolerated Dose and Recommended Phase 2 Dose of TENPA (Targeting-Enhancing Nanoparticles of Paclitaxel) in Patients With Advanced Solid Tumor
Brief Title: Phase I Study of TENPA in Advanced Solid Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Yung-Jue Bang (Other)
Responsible Party: Sponsor-Investigator, Yung-Jue Bang, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H1604-140-758
Record Dates: First submitted 2016-11-27; First posted 2016-12-01 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Advanced Solid Tumor

ARMS (1):
- Phase I (Experimental): Part A, Dose escalation TENPA (Targeting-Enhancing Nanoparticles of Paclitaxel) IV once every 3 weeks (Phase I starting dose 75 mg/m2) Part B, Expansion TENPA (Targeting-Enhancing Nanoparticles of Paclitaxel) IV once every 3 weeks (RP2D dose determined in part A)
  Interventions: Drug: TENPA (Targeting-Enhancing Nanoparticles of Paclitaxel)

INTERVENTIONS:
Drug: TENPA (Targeting-Enhancing Nanoparticles of Paclitaxel) — TENPA IV once every 3 weeks (Phase I starting dose 75 mg/m2)

SUMMARY:
The purpose of this study is to investigate the safety and to determine maximum tolerated dose and recommended phase 2 dose of TENPA (Targeting-Enhancing Nanoparticles of Paclitaxel) in patients with advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for voluntary participation in the trial
2. Twenty years of age or older on the day of signing informed consent
3. Advanced solid tumors with no standard treatment available
4. Evaluable disease or have measurable lesion
5. ECOG performance score of 0 or 1
6. Life expectancy ≥ 12 weeks
7. Adequate organ and marrow function as defined below:

   A. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3) B. Haemoglobin ≥ 8.0 g/dL C. Platelet count ≥ 100 x 109/L (>100,000 per mm3) D. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional ULN E. Serum bilirubin ≤ 2 x institutional upper limit of normal (ULN) F. Serum creatinine ≤ 1.5 mg/dL
8. Adequate heart function A. QT interval corrected for heart rate (QTc) ≤ 480 ms
9. In the opinion of the investigator likely to have the willingness to comply with the study protocol during and after the study period and capable of complying with it
10. Negative serum pregnancy test (β HCG) upon study entry and agree to use contraception

Exclusion Criteria:

1. Uncontrolled CNS metastatic disease (radiographically unstable and symptomatic disease). (note) Subjects with previously treated CNS metastases (surgery or stereotactic brain radiation therapy) that are radiographically stable for at least 4 weeks are permitted to enroll. Subjects should not receive corticosteroids within 3 weeks prior to study enrollment.
2. History of leptomeningeal carcinomatosis; brain metastasis with seizure not controlled with standard medical management.
3. Major surgery within 4 weeks: patient must have recovered from any effects of any major surgery.
4. History of hematopoietic stem cell transplantation or solid organ transplantation
5. History of Gilbert's syndrome
6. Prior malignancy except:

   Basal cell carcinoma and squamous cell carcinoma of the skin that has undergone potentially curative surgery, in situ cervical cancer that has undergone potentially curative surgery and had no evidence of recurrence at least in past 3 years, other malignancy that has undergone curative surgery and had no evidence of disease at least in past 5 years.
7. Significant cardiovascular disease, such as: history of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months; History or current evidence of clinically significant arrhythmia or conduction disorder, except symptomatic congestive heart failure (CHR), atrial fibrillation, and paroxysmal supraventricular tachycardia (PSVT)
8. Sustained uncontrolled hypertension
9. Test results indicating active infection with human immunodeficiency virus (HIR) or hepatitis B or C, defined by positive serology testing (note) inactive hepatitis B carrier on antiviral agents are permitted to enroll.
10. Neuromuscular disorder associated with CK elevation (eg. Inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, and spinobulbar muscular atrophy)
11. Uncontrolled intercurrent illness or symptoms including, but not limited to, ongoing or active infection, bowel obstruction, psychiatric illness/social situations that would limit compliance with study requirement.
12. Radiation therapy within 2 weeks of the first dose of study drug: patient must have recovered from any effects of radiation therapy
13. Pregnant or breast feeding.
14. Female subjects of childbearing potential within the projected duration of the study, starting with the screening visit through 30 days after the last dose of study drug.

    Female of childbearing potential are defined as those who are not surgically sterile (i.3., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or who are not postmenopausal (defined as 12 months with no menses without an alternative medical cause). Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
15. Non-sterilized males who are sexually active with a female partner of child bearing potential from screening through 30 days after receipt of the final dose of study drug.
16. Any medical, psychiatric or cognitive disorder that compromise the ability of the subject to give informed consent, comply with the study protocol, and complete the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | at least one cycle of treatment (3 weeks)
Maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) | at least one cycle of treatment (3 weeks)

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 3 weeks
Area Under the Curve [AUC] | 3 weeks
Response rate (RR) | 6 weeks
Progression-free survival (PFS) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea